CLINICAL TRIAL: NCT01268852
Title: Effectiveness of Insignia ™ Versus Standard Orthodontic Treatment With Damon Q Brackets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Insignia versus Damon Q
Record Dates: First submitted 2010-12-28; First posted 2010-12-31 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2016-01

CONDITIONS: Orthodontic Treatment; Fixed Appliances; Insignia; DamonQ Brackets

STUDY DESIGN:
Intervention Model Description: Compare treatment between two appliance systems
Who Masked: Investigator, Outcomes Assessor
Masking Description: Masking was done with generated cmputer randomisation and sealed opaque enveloppes
Oversight: Data Monitoring Committee: No

ARMS (2):
- Damon (Active Comparator): Standard self ligating orthodontic Damon brackets
  Interventions: Device: Damon self ligating orthodontic bracket
- Insignia (Experimental): Innovative self ligating orthodontic bracket
  Interventions: Device: Insignia self ligating orthodontic bracket

INTERVENTIONS:
Device: Damon self ligating orthodontic bracket — Orthodontic treatment with Damon self ligating bracket
  Arms: Damon
Device: Insignia self ligating orthodontic bracket — Orthodontic treatment with Insignia self ligating bracket
  Arms: Insignia

SUMMARY:
The hypotheses tested in this study are: There is a statistical significant difference, in treatment duration and result of treatment in cases treated using traditional Damon Q brackets or using Insignia.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects, both male and female
* No cleft lip or palate or other craniofacial anomalies
* Treatment with full fixed orthodontic appliances is indicated
* Complete permanent dentition except for upper second and all third molars
* Class I, Class II or Class III first molar relationship )1/2 pb or less off)
* No previous orthodontic treatment
* Age between 12 and 30 years of age
* Study models and lateral cephalograms taken not more than 1 month before selection
* Informed consent signed by patients and parents

Exclusion Criteria:

* Cleft lip and palate and craniofacial anomalies
* Syndromes affecting bone (formation) or teeth
* Agenesis of teeth
* Missing first molars
* No bridges or implants
* Orthognathic cases
* History of periodontal disease
* Intake of drugs affecting tooth movement and/or bone formation
* Pregnancy

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 180 (Actual)
Dates: Start 2011-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Total treatment duration | treatment duration
  duration assesed from start treatment to the removal of appliances

SECONDARY OUTCOMES:
Quality of treatment | at start of treatment wand when finished treatment
  Using one quality grading system: PAR-index
Difference between the planning and the outcome of treatment of the Insignia cases | at start of treatment
  time in minutes with planning the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hero Breuning, Principal Investigator — Radboud university Medical centre Nijmegen, The Netherlands
Locations (1):
- Department of Orthodontics and Craniofacial Biology, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Derived] Penning EW, Peerlings RHJ, Govers JDM, Rischen RJ, Zinad K, Bronkhorst EM, Breuning KH, Kuijpers-Jagtman AM. Orthodontics with Customized versus Noncustomized Appliances: A Randomized Controlled Clinical Trial. J Dent Res. 2017 Dec;96(13):1498-1504. doi: 10.1177/0022034517720913. Epub 2017 Jul 25. PMID 28742420